CLINICAL TRIAL: NCT00936624
Title: A 12 Week, Multi-center,Randomized, Double Blinded, Parallel Group, Placebo-controlled, 4-arm, Dose Finding Trial to Assess the Efficacy and Safety of SOTB07 in Persistent Asthma
Brief Title: Dose Finding Trial to Assess the Efficacy and Safety of SOTB07 in Persistent Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SK Chemicals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SOTB07_AST_II_2008
Record Dates: First submitted 2009-07-08; First posted 2009-07-10 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2013-12

CONDITIONS: Asthma
Keywords: Persistent asthma
MeSH Terms: conditions — Asthma | interventions — montelukast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- SOTB07 100mg (Experimental)
  Interventions: Drug: SOTB07
- SOTB07 200mg (Experimental)
  Interventions: Drug: SOTB07
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo
- Montelukast 10mg (Active Comparator)
  Interventions: Drug: montelukast

INTERVENTIONS:
Drug: SOTB07 — SOTB07 100mg
  Arms: SOTB07 100mg
Drug: SOTB07 — SOTB07 200mg
  Arms: SOTB07 200mg
Drug: placebo — placebo
  Arms: Placebo
Drug: montelukast — montelukast 10mg po, bid, 12week
  Arms: Montelukast 10mg

SUMMARY:
This study is a dose finding trial to assess the efficacy and safety of SOTB07 in persistent asthma.

DETAILED DESCRIPTION:
A 12 week, Multi-center, Randomized, Double blinded, Parallel group, Placebo-controlled, 4-arm, Dose finding trial to Assess the Efficacy and Safety of SOTB07 in persistent asthma.

ELIGIBILITY:
Inclusion Criteria:

1. Male or eligible female subjects aged 15 years or more
2. A female is eligible if she is of:

   * Non-child bearing potential (i.e., physiologically incapable of becoming pregnant), including any female who is at least 2 year after post- menopausal
   * Child bearing potential and agrees to the acceptable contraceptive methods used consistently and correctly
   * Negative pregnancy test at screening
3. Non-smoker for at least 1 year, a pack history of ≤ 10 pack years
4. Symptom of persistent asthma, as defined by the National Institute of Health (NIH)
5. 50% ≤ FEV1 ≤ 85% predicted at screening visit (withholding inhaled, short acting ß-agonist for 6 hours)
6. FEV1 reversibility ≥ 12% and 200 ml at 20-30 minutes after inhalation of a short acting ß-agonist (Salbutamol 2 puffs; 200㎍) at Visit 1 or within 6 months before Visit 1
7. Capable of withholding salbutamol use for ≥ 6 hours prior to clinic visits
8. Appropriately signed and dated informed consent has been obtained

Exclusion Criteria:

1. Active upper or lower respiratory tract infection within 3 weeks before visit 1
2. Emergency room treatment for asthma within 1 month or hospitalization for asthma within 3 months before visit 1
3. Any evidence of infectious, oncologic, or other active pulmonary disease obtained by chest radiography within 12 months before visit 1
4. Clinically significant, in the opinion of the investigator, hematological, liver, renal, heart, neurological disease, or other serious disease
5. Hypersensitivity to any β2-agonist, sympathomimetic drug, leukotriene receptor antagonist or Sophora tonkinensis Radix Rhizoma
6. Clinically significant and uncontrolled psychiatric disease or history of drug or alcohol abuse
7. Inhaled, oral or parenteral corticosteroids within 4 weeks before visit 1
8. Change of Immunotherapy within 6 months before visit 1
9. Administration of the antiasthma agent within 1 week of visit 1
10. Administration of any other medication which may affect the course of asthma, or interact with sympathomimetic amines
11. Participation in study using an experimental medication within 1 month before visit 1
12. Other ineligible subject in the opinion of the investigator

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 245 (Actual)
Dates: Start 2009-07; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
% change from baseline for FEV1 at each visit | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sangheon Cho, professor, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea